CLINICAL TRIAL: NCT01310478
Title: PhaseⅠClinical Study of Recombinant Human Endostatin in Combination With mFOLFOX6 as Initial Therapy for Patients With Metastatic Colorectal Cancer
Brief Title: Recombinant Human Endostatin in Combination With mFOLFOX6 in Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials,Shanghai Cancer Center, Fudan University, Department of medical oncology, Shanghai Cancer Center,Fuandan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIM-85
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2010-06

CONDITIONS: Colorectal Neoplasm
Keywords: Recombinant human endostatin; Metastatic colorectal cancer; DLT; MTD; Pharmacokinetics
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endostar combined with mFOLFOX6 (Experimental)
  Interventions: Drug: recombinant human endostatin (Endostat)

INTERVENTIONS:
Drug: recombinant human endostatin (Endostat) — mFOLFOX6:Oxaliplatin 85 mg/m2 d1 Leucovorin 400 mg/m2 d1+5-FU 400 mg/m2 bolus d1+5-FU 2.4 CIV 46h Endostar 7.5mg/m2/d～45mg/m2/d continous intravenous d4～d14
  Other Names: Endostar

SUMMARY:
To investigate safety and tolerance of dose-escalation of infusional recombinant human endostatin in combination with mFOLFOX6 as initial therapy for patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Recombinant human endostatin(Endostar) is commonly used through intermittent intravenous adminstration in routine clinical practice in China. It is very difficult to maintain steady-state of plasma concentration of this agent due to this manner of application. Continous infusional Endostar was designed to alter the imblance of concentration to avoid compromising efficacy of anti-angionesis therapy.The strategy of dose-escalation was used in this study in order to obtain the optimal dosage of Endostar for the next phase Ⅱ trial.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Histological or cytological confirmed adenocarcinoma of the colon or rectum
3. Age between 18 and 70 years.
4. Patients must have received no prior systemic therapy for metastatic disease. Anyadjuvant/neoadjuvant oxaliplatin therapy must have been received >12 months prior to study entry and adjuvant/neoadjuvant 5-FU must have been received >6 months prior to study entry. Patients who have previously been disease free following a neoadjuvant chemotherapy regimen and resection of all primary tumour and metastatic disease are eligible..
5. ECOG Performance Status of 0 or1
6. Life expectancy of at least 12 weeks
7. The required evidence of measurable lesions should be at least 10 mm in the longest diameter by spiral computed tomography scan or 20 mm with conventional techniques (RECIST criteria)
8. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   * Hemoglobin > 9.0 g/dl
   * Absolute neutrophil count (ANC) >1,500/mm3
   * Platelet count 100,000/μl
   * Total bilirubin < 1.5 times the upper limit of normal ALT and AST < 2.5 x ULN(< 5 x ULN for patients with liver involvement of their cancer)
   * ALP< 4 x ULN
   * PT-INR/PTT < 1.5 x upper limit of normal
   * Serum creatinine < 1.5 x ULN

Exclusion Criteria:

1. History of cardiac disease:

   * congestive heart failure >NYHA class 2
   * with a history of symptomatic coronary artery disease(including angina and myocardial infarction) or other ischemic heart disease
   * cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
2. History of HIV infection or chronic hepatitis B or C (high copy number of HBV).
3. Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
4. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
5. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
6. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma within 5 years.
7. Recent (<28 days) major thoracic or abdominal surgery prior to entry into the studyor a surgical incision that is not fully healed
8. Known hypersensitivity to recombinant human endostatin, oxaliplatin, 5-FU, leucovorin, capecitabine or any of the excipients of these products
9. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
10. Peripheral neuropathy ≥CTC grade 2
11. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
12. Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial (and men for at least 3 months after last administration of study medication).

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity and maximum tolerance dose of continous intravenous Endostar in combination with mFOLFOX6 | 14 days

SECONDARY OUTCOMES:
Parameters of human pharmacokinetics of continous intravenous Endostar in combination with mFOLFOX6 | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China